CLINICAL TRIAL: NCT06063356
Title: Effects of Dextrose Prolotherapy on Pain, Muscle Strength, Proprioception and Quality of Life in Patients With Knee Osteoarthritis: Randomized Controlled Trial
Brief Title: Effects of Dextrose Prolotherapy in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ekin Ilke Sen, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulU-2023-77979112
Record Dates: First submitted 2023-09-19; First posted 2023-10-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose Prolotherapy (Active Comparator): Intra-articular Injection: A total of 5 cc of 25% dextrose solution (4 cc of 30% dextrose + 1 cc of saline) will be administered to the patellofemoral joint space in each patient with the same technique using the supero-lateral technique using a sterile injector with a 20 gauge needle tip.
  Interventions: Procedure: Intra-articular and extra-articular Dextrose Prolotherapy injection; Procedure: Intra-articular and extra-articular Saline injection
- Saline (Active Comparator): Intra-articular Injection: Using a sterile syringe with a 20 gauge needle tip, a total of 5 cc of saline will be administered to the patellofemoral joint space in each patient with the same technique using the supero-lateral technique.
  Interventions: Procedure: Intra-articular and extra-articular Dextrose Prolotherapy injection; Procedure: Intra-articular and extra-articular Saline injection

INTERVENTIONS:
Procedure: Intra-articular and extra-articular Dextrose Prolotherapy injection — In the prolotherapy group, 28 patients will receive intra-articular 5 cc 25% dextrose solution (4 cc 30% dextrose + 1 cc saline) and extra-articular 10 cc 15% dextrose solution (5 cc 30% dextrose + 2.5 cc saline + 2.5 cc 1% lidocaine) in 3 sessions.Extra-articular Injection: Using a sterile syringe with a 27 gauge needle tip (Dental), the points previously found and marked with US (medial collateral ligament, lateral collateral ligament, patellar ligament and adhesion sites of coronary ligaments; pes anserine and superior patellar regions) perpendicular to the surface, using peppering technique, a total of 10 cc of 15% dextrose solution (5 cc 30% dextrose + 2.5 cc saline + 2.5 cc 1% lidocaine) will be injected in small volumes (0.5cc-1cc) at each point.Injection applications will be done at weeks 0 - 3 - 6.
Procedure: Intra-articular and extra-articular Saline injection — In the saline group, 28 patients are planned to receive 3 sessions of intra-articular 5 cc saline and extra-articular 10 cc lidocaine-serum physiologic solution (5 cc saline + 5 cc 1% lidocaine).Injection applications will be done at weeks 0 - 3 - 6.

SUMMARY:
In this prospective, randomized, controlled, single-blinded study, we aimed to evaluate the effects of Dextrose Prolotherapy injections in patients with chronic knee osteoarthritis.

DETAILED DESCRIPTION:
Patients admitted to Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation Outpatient Clinic with a diagnosis of knee osteoarthritis and who meet the inclusion criteria will be included in the study. Patients will be informed verbally and in writing about the purpose, duration and method of the study and will be asked to sign an "Informed Consent Form" after their consent is obtained.

In our study, the investigators aimed to evaluate the effects of dextrose prolotherapy injections in patients with chronic knee osteoarthritis. The duration of the study was determined as 8 months and it was planned to include 33 patients for each group to be randomized by computer program according to the order of application and 66 patients in total.

Patients who meet the inclusion and exclusion criteria will be randomized into 2 groups and the first group will receive Dextrose Prolotherapy and home exercise program and the second group will receive saline injection and home exercise program.

After the application, patients will be questioned in terms of side effects and complications.

History and demographic characteristics such as age, gender, height, weight, marital status, educational level and occupation will be questioned, and medical history such as history of comorbidities and treatment approaches will be determined. In the physical examination, knee tests (ROM measurements, ligament tests, meniscus tests, tests for osteoarthritis) will be performed and TUG (Timed Up and Go) Test will be evaluated. Direct knee radiographs will be evaluated according to Kellgren-Lawrence Gonarthrosis Staging. The average and maximum level of pain during activity, at rest and at night will be questioned with the Visual Analog Scale (0-10 points). WOMAC pain score and WOMAC total scores will be questioned. Isokinetic muscle strength and proprioception will be evaluated with Biodex Isokinetic Dynamometer in our clinic. Functional status will be evaluated with Euro-Qol Quality of Life Scale. The evaluations will be performed by the researcher who is blinded to the applications.

Assessments will be made before treatment, 1 month, 3 months and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral symptomatic knee pain resistant to conservative treatment for at least three months
* Presence of Kellgren-Lawrence stage 2-3 osteoarthritis on current anterior-posterior knee radiographs
* 40-65 years of age
* Functional ambulation scale stage 4-5

Exclusion Criteria:

* Kellgren-Lawrence stage 1 or stage 4 osteoarthritis on current anterior-posterior knee radiographs
* Intra-articular knee injection within the last six months
* History of severe trauma to the knee within the past six months
* Concomitant severe meniscus or ligament injury, surgery applied to the knee area
* Presence of severe effusion, inflammatory joint disease, infection, hematological and oncological disease in the knee.
* Having a bleeding disorder and / or using warfarin
* Patients with hemoglobin less than 11g/dL and platelet count of less than 150,000 platelets per microliter
* Presence of uncontrolled diabetes mellitus
* Presence of cardiac or systemic disease that may affect exercise
* The presence of neurological disease and psychiatric disease such as Parkinson's disease, stroke history that may affect balance
* Body Mass Index ≥35 kg/m²
* Allergy to local anesthetic

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures knee pain, stiffness, and physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for the three subscales gives a total WOMAC score. High scores are associated with more pain, stiffness, and poor function, while low scores indicate well-being.

SECONDARY OUTCOMES:
Change from baseline stiffness and physical function at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures knee pain, stiffness, and physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for the three subscales gives a total WOMAC score. High scores are associated with more pain, stiffness, and poor function, while low scores indicate well-being.
Change from baseline activity pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Activity pain (0-10 point). Higher scores mean a worse outcome
Change from baseline rest pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Rest pain (0-10 point). Higher scores mean a worse outcome
Change from baseline night pain score at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Visual Analogue Scale-Night pain (0-10 point). Higher scores mean a worse outcome
Change from baseline quality of life at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  The EuroQOL (EQ-5D-3L) scale is a scale developed to assess health-related quality of life and consists of two parts. The first part describes the health profile in 5 dimensions (mobility, self-care, social life, pain and psychological state). Each dimension includes 3 statements according to the degree of difficulty (1- some problem; 2-moderate; 3-much problem), the second part includes a visual analog scale (VAS) in which respondents rate their current health status from 0 to 100.
Change from baseline functional balance at 1-months, 3-months and 6-months | Baseline, 1-month, 3-month, 6-month
  Timed Up and Go test requires the person to stand up from a standard chair in which they are sitting, walk 3 m at a comfortable speed to the marked place on the floor, turn around, walk backwards to the starting point and return to the sitting position in the chair. The time taken for the person to complete the test is measured in seconds. The timing of the test is related to the function.
Change from baseline muscle strength and proprioception at 3-months and 6-months | Baseline, 3-month, 6-month
  Isokinetic muscle strength and proprioception will be evaluated with Biodex Isokinetic Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Ekin I Sen, Assoc.Prof., Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)